CLINICAL TRIAL: NCT01100268
Title: Enhancing Attention in Adults With Compulsive Hoarding: A Pilot Study
Brief Title: Enhancing Attention in Adults With Compulsive Hoarding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6133
Record Dates: First submitted 2010-04-05; First posted 2010-04-08 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Hoarding Disorder
Keywords: Hoarding
MeSH Terms: conditions — Hoarding Disorder; Hoarding | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylphenidate ER (Experimental): Subjects will start at 18mg/day; the dose will be increased in increments of 18mg per week to reach 72mg/day.
  Interventions: Drug: Methylphenidate ER

INTERVENTIONS:
Drug: Methylphenidate ER — Subjects will start at 18mg/day; the dose will be increased in increments of 18mg per week to reach 72mg/day.
  Other Names: Concerta

SUMMARY:
Available data suggest that compulsive hoarders have cognitive deficits, particularly with sustaining attention that might contribute their hoarding symptoms.

DETAILED DESCRIPTION:
Compulsive hoarders perform significantly worse than healthy controls on standard attention tasks. These data suggest that the inability to sustain focus may interfere with hoarders' ability to organize, categorize and make decisions about discarding possessions. Stimulants are first-line treatments for ADHD, improve CPT performance in people with ADHD and enhance school performance in children with ADHD. Extended release formulations, such as methylphenidate ER, are associated with better medication compliance. Together, these data suggest that adjunctive methylphenidate ER might be a novel way to improve attention in compulsive hoarders which might improve hoarding symptoms.

The investigators hypothesis is that adjunctive methylphenidate ER will improve attention in compulsive hoarders aged 18-55. The investigators will also explore the safety of methylphenidate ER administration in compulsive hoarders.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant compulsive hoarding (Proposed DSM-V criteria) that is principal (i.e. currently most severe and needing of treatment) and has been present for at least one year.
* At least moderate attentional difficulties.
* Able to provide consent.
* Patients can be on or off of serotonin reuptake inhibitors (SRIs) or serotonin and norepinephrine reuptake inhibitors (SNRIs) but dose must be stable for 12 weeks prior to study.

Exclusion Criteria:

* Currently taking any psychotropic medications other than SRIs or SNRIs.
* Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder or other psychotic disorder.
* Current major depression is permitted if clearly secondary in importance to the hoarding.
* Judged clinically to be at risk of suicide (suicidal ideation, severe depression or other factors)
* Any cardiovascular abnormality that increases the risk of participation, including significant history of cardiovascular disease or family history of sudden death.
* Any medical or neurological disorder that increases the risk of participation or that is a medical contraindication for taking methylphenidate (e.g. glaucoma or Tourette's syndrome).
* Current use of any drug that is contraindicated with methylphenidate (e.g. monoamine oxidase inhibitors).
* Female patients who are pregnant or nursing.
* Current or previous treatment with methylphenidate or CBT for hoarding.
* Current ETOH/drug abuse or dependence disorder of dependency in the past 6 months.
* Individuals with mild cognitive impairments, dementia, or significant intellectual deficits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I. Rodriguez, M.D., Ph.D., Principal Investigator — Columbia-NYSPI-RFMH
Locations (2):
- United States (2):
  - Institute of Living, Hartford, Connecticut
  - New York State Psychiatric Insitute, New York, New York

REFERENCES:
- [Background] Rodriguez CI, Bender J Jr, Morrison S, Mehendru R, Tolin D, Simpson HB. Does extended release methylphenidate help adults with hoarding disorder?: a case series. J Clin Psychopharmacol. 2013 Jun;33(3):444-7. doi: 10.1097/JCP.0b013e318290115e. No abstract available. PMID 23609401
- See also: Columbia University Obsessive-Compulsive Disorder Clinic — http://www.columbia-ocd.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period are: April 2010-July 2010 Location: Outpatient clinic
Period: Overall Study
Arm/Group | Methylphenidate ER
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Individuals with Hoarding Disorder
Arm/Group | Methylphenidate ER
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Met and Exceeded Response Criteria of Attention Deficit Hyperactivity Disorder Symptom Scale
Description: Patients given Attention Deficit Hyperactivity Disorder Symptom Scale (ADHDSS), a measure of the features of Attention Deficit Hyperactivity Disorder including inattention, hyperactivity, and impulsivity. This scale has shown excellent reliability in prior studies of individuals with HD. For the ADHDSS the minimum units are 0 and Maximum units on the total scale are 54 (adult). The higher the number on the ADHDSS, the more severe the symptoms. Response was defined as at least a 30% reduction on the ADHDSS.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Methylphenidate ER
Number analyzed (Participants) | 4
participants | 4

2. Secondary Outcome: Number of Patients Who Met Response Criteria for the Saving Inventory-Revised.
Description: Patients given Saving Inventory-Revised (SI-R), an evidence-based measure of three features of hoarding: excessive acquisition, difficulty discarding, and clutter. For the SI-R the minimum units are 0 and Maximum units on the total scale are 92. The higher the number on the SI-R, the more severe the symptoms. Response was defined as at least a 25% reduction on the SI-R.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Methylphenidate ER
Number analyzed (Participants) | 4
participants | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Methylphenidate ER
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No